CLINICAL TRIAL: NCT06402084
Title: The Relationship Between Fatty Liver and Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Samar Saad Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Samar Saad Abdelrahman, Resident doctor at tropical medicine and gastroenterology Department at sohag univerisity, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-24-04-013MS
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: The Relationship Between Fatty Liver and Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: cases
  Interventions: Diagnostic Test: abdominal ultrasound
- group B: controls
  Interventions: Diagnostic Test: abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: abdominal ultrasound — abdominal ultrasound and lipid profile will be done
  Other Names: lipid profile

SUMMARY:
clinicopathological result of a common is (NAFLD) alcoholic fatty liver disease-nNo 30% of -NAFLD affects 20% .not caused by alcohol intake is chronic liver disease thatsuch as conditions spectrum of population and can be characterized by wide general et Chalasani( steatosis by isolated intracellular fat deposition marked noninflammatory .al., 2012)

homeostasis and egulation of hepatic cholesterol NAFLD occurs due to the dysr . NAFLD is liver in triglycerides and free cholesterol, free fatty acids, accumulation ofabdominal and with insulin resistance, diabetes mellitus, metabolic syndrome associatedimplicated in the be can NAFLD that suggested reports the arge number ofL .obesity kidney diseases as well as cancersf cardiovascular, pulmonary, and pathology o .2015) et al., (Arguello

their course of the Patients with breast cancer commonly develop NAFLD during .45.2%-2.3% approximately cancer is disease. The incidence of NAFLD in breast by influenced metabolic profile and is patient's NAFLD seems to be associated with cardiovascular and resistance insulin causingand treatment, breast cancer complications (Lee et al., 2017).

modulators term estrogen inhibition with selective estrogen receptors-Long liver with tamoxifen fatty incidence of The s been reported to cause NAFLD.ha (SERMs)of NAFLD development in impact heT . use an that for aromatase inhibitoruse is higher th et al., (Yang breast cancer patients after hormonal treatment has not yet been elucidated .)6201

main and is aworldwide most common cancer in womenBreast cancer is the decreasing with has been cancer breast from ityortalM .women in death cancer of causeIt is well known time given the advances in screening strategies and adjuvant treatments. incidence of breast cancer is correlated with age and other risk factors such asthat the mutation, family history of )BRCA2( breast cancer gene2 or )BRCA1(gene1breast cancer al.,et Berry( and hormonal factors chest the to breast cancer, therapeutic radiation5).200

Breast cancer is divided according to the hormone receptors into either hormone receptor-positive tumors which are estrogen receptor-positive (ER-positive) and progesterone receptor-positive (PR-positive). These tumors express hormone receptors. This means they have a lot of hormone receptors. Hormone receptor-negative tumors are estrogen receptor-negative (ER-negative) and progesterone receptor-negative (PR-negative). These tumors donot express hormone receptors. This means they have few or no hormone receptors. About 70% to 80% of newly diagnosed breast cancers are hormone receptor- .al., 2017) (Wang et positive

ELIGIBILITY:
Inclusion Criteria:

* 65 years old)-Age (18-1

performance (PS0;full active,noPerformance status < or equal to 2 Patients with-2PS1;strenuous physical activity restricted,fully ambulatory and able to ----restriction.care but unable to carry out any work -PS2;capable of all self-------carry out light work.activities up and about >50% of woking hours)

Exclusion Criteria:

* Patients who had double malignancy.-1

Patients who had severe comorbidities -2

heart failure…..etc,)(pulmonary failure,Renal failure,

Those who declined cancer treatment before completing 85% of the planned dosage -3 hose who are lost during the follow up period.tor

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: breast cancer patients will be included,Patients who were recently diagnosed as breast cancer patients will be included,examined and their files will be studied.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
lipid profile in patients with breast cancer | 1 year
  The relationship between Fatty Liver and Breast Cancer by abdominal ultrasound and lipid

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ; American Gastroenterological Association; American Association for the Study of Liver Diseases; American College of Gastroenterologyh. The diagnosis and management of non-alcoholic fatty liver disease: practice guideline by the American Gastroenterological Association, American Association for the Study of Liver Diseases, and American College of Gastroenterology. Gastroenterology. 2012 Jun;142(7):1592-609. doi: 10.1053/j.gastro.2012.04.001. Epub 2012 May 15. No abstract available. PMID 22656328
- [Background] Arguello G, Balboa E, Arrese M, Zanlungo S. Recent insights on the role of cholesterol in non-alcoholic fatty liver disease. Biochim Biophys Acta. 2015 Sep;1852(9):1765-78. doi: 10.1016/j.bbadis.2015.05.015. Epub 2015 May 29. PMID 26027904
- [Background] Yang YJ, Kim KM, An JH, Lee DB, Shim JH, Lim YS, Lee HC, Lee YS, Ahn JH, Jung KH, Kim SB. Clinical significance of fatty liver disease induced by tamoxifen and toremifene in breast cancer patients. Breast. 2016 Aug;28:67-72. doi: 10.1016/j.breast.2016.04.017. Epub 2016 May 27. PMID 27240168
- [Background] Lee S, Jung Y, Bae Y, Yun SP, Kim S, Jo H, Seo HI. Prevalence and risk factors of nonalcoholic fatty liver disease in breast cancer patients. Tumori. 2017 Mar 24;103(2):187-192. doi: 10.5301/tj.5000536. Epub 2016 Aug 24. PMID 27647227